CLINICAL TRIAL: NCT03832465
Title: Visiting Staff, Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan
Brief Title: Intraluminal Mono-antibiotic Therapy for Helicobacter Pylori Infection - A Comparison of Levofloxacin Powder and Levofloxacin Solution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tai-cherng Liou, MD, Principle investigator, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18MMHIS168
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Levofloxacin; Amoxicillin; Proton pump inhibitor; Helicobacter Pylori

STUDY DESIGN:
Intervention Model Description: 50 participants are randomly assigned to receive intraluminal eradication of H. pylori.
  with medicaments containing levofloxacin powder or levofloxacin solution. Patients failed to achieve intraluminal eradication of H. pylori will be randomly assigned to 7-day or 14-day levofloxacin-containing triple therapy (levofloxacin 500 mg once daily, amoxicillin 1 g twice daily, and esomeprazole 40 mg twice daily).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraluminal Levofloxacin powder therapy (Experimental): Group A Crashed powder of film-coated Levofloxacin Tablet (1 gm) for the Intraluminal therapy
  Interventions: Drug: Levofloxacin film-coated tablet
- Intraluminal Levofloxacin solution therapy (Active Comparator): Group B Intravenous solution of Levofloxacin (1 gm) for the Intraluminal therapy
  Interventions: Drug: Levofloxacin intravenous solution

INTERVENTIONS:
Drug: Levofloxacin film-coated tablet — 50 participants are randomly assigned to receive intraluminal eradication of H. pylori.
  with medicaments containing levofloxacin powder or levofloxacin solution.
  Other Names: Leflodal film-coated tablet
  Arms: Intraluminal Levofloxacin powder therapy
Drug: Levofloxacin intravenous solution — 50 participants are randomly assigned to receive intraluminal eradication of H. pylori.
  with medicaments containing levofloxacin powder or levofloxacin solution.
  Other Names: Cravit intravenous solution
  Arms: Intraluminal Levofloxacin solution therapy

SUMMARY:
Helicobacter pylori (H. pylori) is an important causal factor of chronic gastritis, peptic ulcer disease, gastric cancer and gastric lymphoma. The World Health Organization classified H. pylori as a Group 1 carcinogen in 1994. Endoscopic examination is indicated to confirm the above diagnosis for patient with H. pylori infection. The eradication of H. pylori can reduce the recurrence rate of peptic ulcer disease and even has the potential to prevent gastric cancer. H. pylori is the most common chronic bacterial infection in humans. The prevalence of H. pylori is about 30-50% in the Western adult population. It is estimated that about 50% of people are infected with this bacterium in Taiwan.

Triple therapy which contains a proton pump inhibitor and two antibiotics among clarithromycin, amoxicillin, and metronidazole is the most commonly used regimen for H. pylori eradication. The treatment duration is 7 to 14 days. However, the eradication rate of standard triple therapy has fallen below 80% in many countries due to the worldwide increasing prevalence of antibiotic resistant strains.

Several strategies have been proposed to increase the eradication rate in the first line therapy or as a rescue therapy, including extending the treatment duration to 14 days, increasing the doses of antibiotics, the use of four or even five drugs regimen (sequential, concomitant, quadruple or quintuple therapy), and other antibiotics such as levofloxacin. However, these therapies may increase the side effects and costs of treatment, decrease the compliance of patients and increase the rate of worldwide antibiotic resistance steadily. The WHO has listed H. Pylori as one of 16 antibiotic-resistant bacteria that have the greatest threat to human health in February, 2017.

The most commonly used oral antibiotics for the treatment of H. pylori are Amoxicillin、Clarithromycin、Metronidazole、Levofloxacin and Tetracycline.

However, with the increasing rates of antibiotic-resistance for Clarithromycin and Metronidazole, the Clarithromycin and Metronidazole were replaced by Levofloxacin as a first line or second line treatment in some area. However, the eradication rate of Levofloxacin-containing triple therapy is suboptimal in many countries. The investigators aim to compare the efficacy of different formulation between Levofloxacin Powder and Levofloxacin Solution in the Intraluminal levofloxacin therapy, and to improve the eradication efficacy of one-week Levofloxacin-containing triple therapy via the Intraluminal therapy.

DETAILED DESCRIPTION:
During the endoscopic examination, patient is sedated with intravenous Dormicum 5mg (5mg/1ml/amp), the vital signs will be closely monitored by physiological monitor (PHILIPS SureSigns VM6). The treatment will be terminated immediately if unstable vital sign detected or if patient asks for termination. Patients will receive tests to evaluate H. pylori colonization in the gastric cardia (UFT300) and duodenal bulb (CLO). With endoscope apparatus, the gastric mucus is irrigated with acetylcysteine solution and the pH value of gastric juice will be measured with the pH test strips before irrigation and after irrigation.

The investigators randomly assigned medicaments containing different formulation (powder or solution ) of levofloxacin to dispense on the surface of gastric mucosa and duodenal mucosa of duodenal bulb. After the intraluminal therapy, patients will rest for 30 to 60 minutes and go home if the effect of sedation subsided. Patients can take meal if no abdominal discomfort. C13-Urea breath test (UBT) will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy. Patients failed to achieve intraluminal eradication of H. pylori will be randomly assigned to 7-day or 14-day levofloxacin-containing triple therapy (levofloxacin 500 mg once daily, amoxicillin 1 g twice daily, and esomeprazole 40 mg twice daily). The C13-UBT will be used to assess the existence of H. pylori 6 weeks after the oral antibiotic therapy. The overall eradication rates of the intraluminal therapy plus the oral antibiotics therapies will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 years and 75 years
2. Patients have H. pylori infection and have not treated with oral antibiotics
3. Patients are willing to receive the intraluminal therapy. The written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

1. Children and teenagers aged less than 20 years or adult greater than 75 years
2. Contraindication for endoscopic examination or food retention in the gastric lumen.
3. History of gastrectomy; Gastroduodenal stenosis、deformity or obstruction; Gastroduodenal malignancy, including adenocarcinoma and lymphoma
4. Contraindication to treatment drugs: previous allergic reaction to Proton pump inhibitors, Amoxicillin, Levofloxacin, Acetylcystein, and pregnant or lactating women
5. Severe concurrent acute or chronic illness: renal failure, decompensated cirrhosis of liver, incurable malignant disease
6. Patients who cannot give informed consent by himself or herself.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
Eradication rate of the intraluminal Levofloxacin therapy | C13-UBT will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy.
  A Comparison of different formulation between Levofloxacin Powder and Levofloxacin solution

SECONDARY OUTCOMES:
Incidence of adverse effects of the intraluminal Levofloxacin therapy | within 7 days after finishing the intraluminal therapies
  A Comparison of different formulation between Levofloxacin Powder and Levofloxacin solution
Eradication rates of 7-day or 14-day levofloxacin-containing triple therapy | C13-UBT will be used to assess the existence of H. pylori 6 weeks after the levofloxacin-containing triple herapies.
  A Comparison of the eradication rates of 7-day or 14-day levofloxacin-containing triple therapy after intraluminal therapy
The overall eradication rate | 3-6 months after finishing the intraluminal therapy
  The overall eradication rates of the intraluminal therapy plus oral antibiotics therapies were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-cherng Liou, MD, Principal Investigator — Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital
Locations (1):
- Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan, Taipei, Taiwan